CLINICAL TRIAL: NCT02788773
Title: A Phase II Study of Durvalumab (MEDI4736) With or Without Tremelimumab in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Durvalumab With or Without Tremelimumab in Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I232
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Durvalumab plus Tremelimumab (Experimental): Durvalumab-IV for 60 minutes day 1 every 4 weeks Tremelimumab-IV every 60 minutes day 1, cycles 1-4
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Arm B - Durvalumab alone (Experimental): Durvalumab-IV for 60 minutes day 1 every 4 weeks
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab
Drug: Tremelimumab
  Arms: Arm A - Durvalumab plus Tremelimumab

SUMMARY:
The purpose of this study is to find out the effects of giving durvalumab alone or in combination with tremelimumab on this type of cancer. In addition, this study will look at the side effects of durvalumab when given alone or in combination with tremelimumab.

DETAILED DESCRIPTION:
Durvalumab is a new type of drug for many types of cancer. Laboratory tests show that it works by allowing the immune system to detect cancer and stimulate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals and has been studied in nearly 2000 people and seems promising but it is not clear if it can offer better results than standard treatment alone.

Tremelimumab is a new type of drug for various types of cancers. It works in a similar way to durvalumab and may improve the effect of durvalumab. This may also help slow the growth of the cancer cells or may cause cancer cells to die. Tremelimumab has been shown to shrink tumours in animals and has been studied in nearly 1500 people and seems promising but it is not clear if it can offer better results than standard treatment alone when used with durvalumab

Combinations of durvalumab and tremelimumab have also been studied and when combined have been shown to increase tumour shrinkage in animals compared to either drug alone. While the combination has been studied in 217 people, it is not clear if it can offer better results than standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the prostate that is castrate resistant.
* Disease progression as defined as one or both of the following: PSA Progression: A rising PSA with 2 subsequent rises over a reference value (not necessarily consecutively), measured a minimum of one week apart. The PSA that confirms progression must have a value of ≥ 2 ng/ml (ug/L).

OR Objective Progression:

* RECIST 1.1
* PCWG 3 Criteria for bone progression
* Patients must be surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 1.7 nM). Patients who have not undergone orchiectomy must continue (or restart if previously discontinued) LHRH therapy throughout the study.
* All patients must have a tumour block from their primary or metastatic tumour available and consent to release the block/recently cut slides for correlative analyses and the centre/pathologist must have agreed to the submission of the specimen(s). The site of planned biopsy must not be the measurable lesion.
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative).
* All patients must have at least one measurable lesion as defined by RECIST 1.1 that has not been the site of the protocol mandated biopsy. The criteria for defining measurable disease are as follows: CT scan (with slice thickness of 5 mm) ≥ 10 mm --> longest diameter; Lymph nodes by CT scan ≥ 15 mm --> measured in short axis
* Patients must be ≥ 18 years of age.
* ECOG performance status 0 or 1.
* Prior Therapy

Systemic Therapy:

0-1 prior regimen of cytotoxic chemotherapy in the CRPC setting is permitted.

Hormonal Therapy:

* Patients must be castrate resistant.
* Have failed/progressed on prior abiraterone and/or enzalutamide.
* Patients must have discontinued anti-androgens for at least 4 weeks prior to study entry (at least 6 weeks for bicalutamide).

Other therapy:

Prior treatment with other agents, such as tyrosine kinase or other targeted agents is permissible.

* Systemic corticosteroids are permitted at a dose equivalent to ≤10 mg prednisone daily and are only permitted for reasons other than prostate cancer treatment (ex: fatigue, anorexia, etc); topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are permitted.
* Bisphosphonates/denosumab are permitted for treatment of hypercalcemia, osteoporosis and skeletal-related events.

Immunotherapy:

Patients may not have received prior immune check point inhibitors (anti PDL1 and anti CTL-4). Vaccines and treatment with oncolytic viruses is permissible.

Patients must have recovered from all reversible toxicity related to prior systemic therapy (chemotherapy and hormone) and have adequate washout as follows:

Longest of one of the following:

* Two weeks;
* The longer of 30 days or 5 half-lives for investigational agents;
* Standard cycle length of standard therapies.

Radiation:

Prior external beam radiation or radium-223 is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and the date of randomization. Exceptions may be made for low-dose non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted. Prior strontium-89 at any time is not permitted

Prior Surgery:

Prior major surgery is permitted provided that a minimum of 28 days (4 weeks) have elapsed between any major surgery and date of randomization, and that wound healing has occurred.

* Laboratory Requirements (Must be done within 7 days prior to randomization):

Abs Neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 90 g/L Bilirubin ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN ≤ 5.0 ULN (if patient has liver mets) Serum Creatinine < 1.25 x ULN or Creatinine clearance ≥ 40mL/min

* Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use male condom plus spermicide while on study and for 6 months after the last dose of durvalumab and tremelimumab, or for 3 months after the last dose of durvalumab alone. Female partners of a male subject must use a highly effective method of contraception throughout this period.
* Male patients should also refrain from donating sperm during the study and for 6 months after the last dose of durvalumab and tremelimumab or for 3 months after the last dose of durvalumab alone.
* Subjects should not donate blood while participating in this study, or for at least 90 days following the last infusion of durvalumab or tremelimumab.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate. Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. The patient's city of residence may be required to verify their geographical proximity. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the tretment, adverse events, and follow-up.
* Patients must agree to return to their primary care facility for any adverse events which may occur through the course of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies requiring concurrent anticancer therapy.
* Patients with brain metastases are not eligible.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia.
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years).
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.
* Live attenuated vaccination administered within 30 days prior to randomization or within 30 days of receiving durvalumab.
* History of hypersensitivity to durvalumab or tremelimumab or any excipient. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, should have a LVEF ≥ 50%.
* Concurrent treatment with other investigational drugs or anti-cancer therapy (except LHRH in patients not surgically castrated).
* Patients with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol (including corticosteroid administration), or would put the patient at risk. This includes but is not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) or tuberculosis or any infection requiring systemic therapy).
  * Active peptic ulcer disease or gastritis.
  * Pneumonitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON Canada; Eric W Winquist, Study Chair — London Regional Cancer Program, London ON Canada
Locations (11):
- Canada (11):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Winquist E, Hotte SJ, Chi K, Sridhar S, Ellard S, Ong M, Iqbal N, Salim M, Emmenegger U, Gingerich JR, Lalani AK, Major P, Kollmannsberger C, Yip S, Hansen A, Finch D, Canil C, Hutchenreuther J, Vera-Badillo F, Smoragiewicz M, Cabanero M, Tsao MS, Ritch E, Wyatt AW, Seymour L. Randomized Phase II Study of Durvalumab with or without Tremelimumab in Patients with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2025 Jan 6;31(1):45-55. doi: 10.1158/1078-0432.CCR-24-1612. PMID 39513948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 15, 2016 to October 1, 2019 from cancer centers in Canada.
Pre-assignment Details: Participants were randomized to one of two treatment arms after assessment of eligibility.
Groups:
- Arm A - Durvalumab Plus Tremelimumab: Durvalumab-IV for 60 minutes day 1 every 4 weeks Tremelimumab-IV every 60 minutes day 1, cycles 1-4
  Durvalumab
  Tremelimumab
- Arm B - Durvalumab Alone: Durvalumab-IV for 60 minutes day 1 every 4 weeks
  Durvalumab
Period: Overall Study
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
Started | 39 | 13
Completed | 39 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone | Total
Number analyzed (Participants) | 39 | 13 | 52
Age, Continuous [Median (Full Range); unit: years] | 72 [52 to 83] | 65 [50 to 83] | 70 [50 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 13 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 34 | 11 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 13 | 52
Baseline PSA (prostate-specific antigen) level [Count of Participants; unit: Participants]
  Higher than or equal to 2 ng/mL but less than 20 ng/mL | 2 | 2 | 4
  Higher than or equal to 20 ng/mL but less than 100 ng/mL | 18 | 4 | 22
  Higher than or equal to 100 ng/mL | 19 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Measured by RECIST 1.1
Description: Response evaluated using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) for target and non-target lesions and assessed by CT or MRI: Complete Response (CR), disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, or in the case of complete remission of the target lesions, when one or more non-target lesions can still be distinguished; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
Number analyzed (Participants) | 39 | 13
Participants | 7 | 0

2. Primary Outcome: Objective Response Rate by iRECIST
Description: Response evaluated using iRECIST (modified Response Evaluation Criteria in Solid Tumours 1.1 for immune-based therapeutics) for target and non-target lesions and assessed by CT or MRI: Complete Response (CR), disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, or in the case of complete remission of the target lesions, when one or more non-target lesions can still be distinguished; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: All patients enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
Number analyzed (Participants) | 39 | 13
Participants | 7 | 0

3. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: A PSA response is defined as 50% fall in PSA from baseline maintained for ≥ 4 weeks, and without evidence of disease progression documented at time of confirmatory values.
Time Frame: 2 years
Population: All patients enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
Number analyzed (Participants) | 39 | 13
Participants | 7 | 0

4. Secondary Outcome: Time to Objective Disease Progression
Description: Time from randomization to objective disease progression documented based on RECIST (Response Evaluation Criteria in Solid Tumours) 1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Population: All patients enrolled
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
Number analyzed (Participants) | 39 | 13
months | 2.79 [2.63 to 3.19] | 2.83 [1.97 to 2.83]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm A - Durvalumab Plus Tremelimumab | Arm B - Durvalumab Alone
All-Cause Mortality (participants affected / at risk) | 34/39 | 12/13
Serious Adverse Events (participants affected / at risk) | 20/39 | 5/13
Other Adverse Events (participants affected / at risk) | 38/39 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Durvalumab Plus Tremelimumab (N=39) | Arm B - Durvalumab Alone (N=13)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Edema limbs (General disorders) | 0 | 1
Edema trunk (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Other immune system disorders (Immune system disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 2 | 1
Confusion (Psychiatric disorders) | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphedema (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Durvalumab Plus Tremelimumab (N=39) | Arm B - Durvalumab Alone (N=13)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 0
Cushingoid (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 4 | 1
Blurred vision (Eye disorders) | 2 | 2
Dry eye (Eye disorders) | 1 | 2
Watering eyes (Eye disorders) | 2 | 0
Other eye disorders (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 2
Constipation (Gastrointestinal disorders) | 17 | 8
Diarrhea (Gastrointestinal disorders) | 14 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 19 | 5
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 14 | 4
Other gastrointestinal disorders (Gastrointestinal disorders) | 2 | 1
Chills (General disorders) | 2 | 1
Edema limbs (General disorders) | 18 | 7
Fatigue (General disorders) | 35 | 11
Flu like symptoms (General disorders) | 4 | 3
Malaise (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 10 | 2
Other general disorders, administration site conditions (General disorders) | 1 | 1
Lip infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 4 | 0
Upper respiratory infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 4 | 1
Other infections and infestations (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 24 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 6
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 3 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 2
Paresthesia (Nervous system disorders) | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 2
Seizure (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 2 | 0
Confusion (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Hematuria (Renal and urinary disorders) | 9 | 2
Urinary retention (Renal and urinary disorders) | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Other renal and urinary disorders (Renal and urinary disorders) | 3 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 | 1
Hot flashes (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Lymphedema (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT02788773/Prot_SAP_000.pdf